CLINICAL TRIAL: NCT03366675
Title: Phase II, Single-arm Study of AZD 2811 Monotherapy in Relapsed Small Cell Lung Cancer Patients [SUKSES-N3]
Brief Title: AZD 2811 Monotherapy in Relapsed Small Cell Lung Cancer Patients [SUKSES-N3]
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early detection of the purpose of the study.
Sponsor: Samsung Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Keunchil Park, Principal Investigator, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-10-071
Record Dates: First submitted 2017-11-27; First posted 2017-12-08 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-02

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — AZD2811

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- AZD2811 (Experimental): AZD2811 200mg IV QD CnD1 & D4 every 4weeks
  Interventions: Drug: AZD2811

INTERVENTIONS:
Drug: AZD2811 — AZD2811 100mg/vial

SUMMARY:
This study is a single arm, multi-center phase II study of AZD 2811 monotherapy in patients with relapsed small cell lung cancer (SCLC) as a second or third line therapy.

Patients will continue to receive study treatment as described above, until they demonstrate objective disease progression (determined by RECIST 1.1) or they meet any other discontinuation criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of fully informed consent prior to any study specific procedures.
2. Patients must be ≥20 years of age.
3. Small cell lung cancer(SCLC) that has progressed during or after first-line therapy.

   * The 1st line regimen must have contained platinum based regimen.
   * Refractory to first-line chemotherapy or relapse within 6 months since the last dose of first-line chemotherapy
   * If the patient correspond to sensitive relapse (relapse more than 6 months since the last dose of first-line chemotherapy), she/he should get second-line treatment.
4. Provision of tumor sample (from either archival or fresh biopsy)
5. Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
6. ECOG performance status of 0-2
7. Patients must have a life expectancy ≥ 3 months from proposed first dose date.
8. Patients must have acceptable bone marrow, liver and renal function measured within 28days prior to administration of study treatment as defined below:

   * Haemoglobin > 9.0 g/dL
   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * White blood cells (WBC) ≥ 3 x 109/L
   * Platelet count ≥100 x 109/L
   * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) except for subject with liver metastases for whom total bilirubin is ≤ 3 x ULN
   * AST(SGOT)/ALT(SGPT) ≤ 2.5 x institutional upper limit of normal(ULN) except for subject with liver metastases for whom AST(SGOT)/ALT(SGPT) is ≤ 5x ULN
   * Alkaline phosphatase(ALP) ≤ 2.5 x institutional upper limit of normal(ULN) except for subject with liver metastases for whom ALP is ≤ 5 x ULN. ALP is not exclusionary if due to the presence of bone metastasis and liver function is otherwise considered adequate in the investigator's judgement.
   * Patients must have creatinine clearance estimated using the Cockcroft-Gault equation of ≥51 mL/min:

   Estimated creatinine clearance = (140-age [years]) x weight (kg) (x F)a serum creatinine (mg/dL) x 72 a where F=0.85 for females and F=1 for males.

   - Albumin ≥ 33g/L
9. At least one measurable lesion that can be accurately assessed by imaging or physical examination.
10. Evidence of non-childbearing status for women of childbearing potential: A woman of childbearing potential must have a negative or urine pregnancy test at screening and confirmed prior to treatment on Cycle 1 Day 1
11. Female patients who are not of childbearing potential and fertile female patients of childbearing potential who agree to use adequate contraceptive measures, who are not breastfeeding. Fertile female patients of childbearing potential should use enhanced methods of contraception from the time of screening until 6 months after discontinuing study treatment. Acceptable methods of contraception include: combined oral or transdermal contraceptives, copper-banded intra-uterine devices and vasectomised partner. All methods of contraception (with the exception of total abstinence) should be used in combination with the use of a condom by their male sexual partner for intercourse. Male patients should be asked to avoid unprotected sex with all sexual partners (by use of condoms) during the study, and for a washout period of 6 months after the last dose of study drug. Where a sexual partner of a male participant is a fertile female patient of childbearing potential, patients should avoid procreation for 6 months after completion of study drug treatment. Patients should refrain from donating sperm from the start of dosing until 6 months after discontinuing study treatment. If male patients wish to father children they should be advised to arrange for freezing of sperm samples prior to the start of study treatment

Exclusion Criteria:

1. Previous enrolment in the present study
2. More than two prior chemotherapy regimen for the treatment of small cell lung cancer
3. Previous treatment with Alisertib
4. Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for >2 years.
5. Treatment with any investigational product during the last 14 days before the enrollment (or a longer period depending on the defined characteristics of the agents used).
6. Patients receiving any systemic chemotherapy, radiotherapy (except for palliative reasons), within 2 weeks from the last dose prior to study treatment The patient can receive a stable dose of bisphosphonates or denosumab for bone metastases, before and during the study as long as these were started at least 4 weeks prior to treatment.
7. Patient has had prescription or non-prescription drugs or other products known to be strong inhibitors/inducers of CYP3A4 which cannot be discontinued prior to Day 1 of dosing and withheld throughout the study until 2 weeks after the last dose of study drug. Washout periods vary between 1 to 5 weeks depending on the medication.
8. With the exception of alopecia, any ongoing toxicities (>CTCAE 4.03 grade 1) caused by previous cancer therapy.
9. Intestinal obstruction or CTCAE 4.03 grade 3 or grade 4 upper GI bleeding within 4 weeks before the enrollment.
10. Resting ECG with measurable QTc > 470 msec on 3 or more time points within a 24 hour period or any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, immediate family history of long QT syndrome or unexplained sudden death under 40 years of age.
11. Patients with cardiac problem as follows: unstable angina pectoris, congestive heart failure, acute myocardial infarction, conduction abnormality not controlled with pacemaker or medication, significant ventricular or supraventricular arrhythmias (patients with chronic rate controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible).
12. Patients at risk of brain perfusion problems(e.g., carotid stenosis hypotension, including a fall in blood pressure of >20mm Hg)
13. Uncontrolled hypertension requiring clinical intervention.
14. Female patients who are breast-feeding or child-bearing
15. Any evidence of severe or uncontrolled systemic disease, active infection, active bleeding diatheses or renal transplant, including any patient known to have human immunodeficiency virus (HIV), active hepatitis B or active hepatitis C
16. Major surgical procedures ≤28 days of beginning study treatment, or minor surgical procedures ≤7 days
17. Known malignant central nervous system (CNS) disease other than neurologically stable, treated brain metastases - defined as metastasis having no evidence of progression or haemorrhage for at least 2 weeks after treatment (including brain radiotherapy).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-10-29 (Actual)

PRIMARY OUTCOMES:
Objective reponse rate (ORR) by RECIST 1.1 | up to 18months
  Assessments to be performed using CT or MRI scans. To be measured

SECONDARY OUTCOMES:
Duration of response | up to 18months
  Assessments to be performed using CT or MRI scans. To be measured
Disease control rate | At 8 weeks
  Assessments to be performed using CT or MRI scans. To be measured
Overall survival(OS) | up to 18 months
  Kaplan-Meier method
Progression-free survival(PFS) | up to 18 months
  Kaplan-Meier method

OTHER OUTCOMES:
Number of participants with Adverse Events as Assessed by CTCAE v4.03 | up to 18months
  CTCAE v4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical center, Seoul, South Korea